CLINICAL TRIAL: NCT00975689
Title: Biomarker Validation for Niemann-Pick Disease, Type C: Safety and Efficacy of N-Acetyl Cysteine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Oxford (Other); Washington University School of Medicine (Other); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 090185; 09-CH-0185
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-04

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: Niemann-Pick Disease, Type C; Biomarkers; N-Acetyl Cysteine; Oxidized Cholesterol; Neurodegeneration; NPC
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Nerve Degeneration | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: N-Acetyl Cysteine — 900mg effervescent tablet; Dosed as 15 mg/kg/day (maximum dose 900 mg per day) for one week, advanced to 30 mg/kg/day (maximum dose 1800 mg per day) for the second week, and then advanced to 60 mg/kg/day (maximum dose 2700 mg) for the remainder of the trial (6 additional weeks).

SUMMARY:
Background:

* Niemann-Pick disease type C (NPC) is a genetic disorder that results in progressive loss of nervous system function by affecting the membranes of nerve cells. There is no known cure for NPC.
* N-acetyl cysteine (NAC) is a drug that has been approved by the Food and Drug Administration to use either orally or IV for the treatment of acetaminophen (Tylenol) poisoning or as an aerosol to reduce the stickiness of mucous in patients with cystic fibrosis. In the body, NAC is converted to an amino acid called cysteine, which cells can convert to a chemical called glutathione. Glutathione is important in helping cells deal with oxidative stress. Based on a number of experiments in cells, mice and patients with NPC, we believe that oxidative stress is increased in NPC. If we can increase glutathione levels, we may be able to decrease the oxidative stress.

Objectives:

- To test the safety and effectiveness of N-acetyl cysteine to treat Niemann-Pick disease (type C).

Eligibility:

- Individuals at least 1 year of age who have been diagnosed with NPC.

Design:

* Patients entering this study will be seen at the National Institutes of Health Clinical Center four times during the 20 weeks of the study. These admissions will occur at the start of the study and at weeks 8, 12, and 20. The first NIH visit will last 2 days, and the other visits will last 1 day.
* Patients will participate in a two-stage study: a period of 8 weeks receiving NAC and a second period of 8 weeks when receiving a placebo (a pill without NAC). Every patient participating in this study will receive NAC during one of the two time periods.
* The two treatment periods will be separated by a wash-out period, 4 weeks when patients will receive neither NAC nor placebo. Patients will also have a 4-week wash-out period at the beginning of the study. Most physician-prescribed medications, such as seizure medications, will be allowed.
* During each visit, examinations, procedures, and tests will be done, including blood and urine samples.

DETAILED DESCRIPTION:
Niemann-Pick Disease, type C (NPC) is an autosomal recessive lysosomal storage disease with progressive neurodegeneration. It is characterized by intracellular accumulation of cholesterol and glycosphingolipids. The age of onset is variable with cases manifesting from infancy to adulthood. Classically, initial neurological symptoms are observed in early to late childhood. Symptoms and signs of NPC include prolonged neonatal jaundice, splenomegaly, and various neurological manifestations, especially ataxia, dysmetria, dysarthria, vertical supranuclear gaze palsy and cognitive decline. Currently there are no approved therapies for NPC. A recent controlled study and a series of case reports suggest some efficacy for miglustat. Miglustat inhibits the biosynthesis of glycosphingolipids. The pathophysiological processes contributing to neurodegeneration in NPC have been intensively studied in NPC mouse models. Potential pathological processes include toxic effects of cholesterol or glycosphingolipid accumulation, deficient oxysterol production, peroxisomal dysfunction, mitochondrial dysfunction, perturbed intracellular calcium homeostasis, inflammation, induction of apoptosis, deficient neurosteroid synthesis, and increased oxidative stress. The degree to which each of these pathological processes contributes to the pathology of NPC is not known; however, the multiple processes involved suggest that combinatorial therapy addressing various aspects of this disorder will be necessary. A major impediment to the development of clinical trials for NPC has been the prior lack of outcome measures. Identifying biomarkers was a major goal of our NPC natural history trial (06-CH-0186). We now have identified multiple biochemical abnormalities in our cohort of patients that may prove useful as biomarkers in a therapeutic trial. The next step is to attempt to validate these potential biomarkers in a therapeutic trial. Thus in this protocol we plan to evaluate the safety and efficacy of N-acetylcysteine to improve a group of biomarkers related to increased oxidative stress.

The goals of this protocol are:

1. To validate the use of biomarkers in a therapeutic trial for NPC.
2. To evaluate the safety of N-acetylcysteine in NPC patients.
3. To evaluate the efficacy of N-acetylcysteine to improve biomarkers associated with increased oxidative stress in NPC patients.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

All patients with an established diagnosis of NPC will be considered for this study. The diagnosis may be based upon either molecular or biochemical testing.

INCLUSION CRITERIA:

1. Diagnosis of NPC by cellular assay or molecular testing.
2. Twelve months of age or older and weight greater than 10 kg.
3. Patient must be able to take the study medication orally or per gastrostomy tube.

EXCLUSION CRITERIA:

1. Patients will be excluded if they cannot travel to the NIH because of their medical condition or are too ill to be cared for at home.
2. Patients will be excluded if they are unable to tolerate the study procedures.
3. Patients will be excluded if they are pregnant (a negative urine pregnancy test will be required for any menstruating female before participation in this study and at each NIH Clinical Center admission). If sexually active, contraception must be used for the duration of the study.
4. Patients will be excluded if they have had prior allergic or hypersensitivity symptoms associated with NAC use.
5. Patients will be excluded from the study if they are unwilling to discontinue the following drugs and supplements for the duration of the study.

   * a. All dietary supplements
   * b. Any antioxidant supplement other than prescribed by the study. This will include dietary juices or drinks being marketed as a source of antioxidants
   * c. CoQ10 supplements
   * d. Any over-the-counter medication being used on a daily basis for which there is not a defined clinical reason
   * e. NAC use
6. Physician prescribed medications will be reviewed on a case-by-case basis. Patients may be excluded if medical therapies could interfere with the study endpoints. Except for carbamazepine, seizure control medications will be allowed. Patients will be excluded if taking carbamazepine or nitroglycerin.
7. Over-the-counter medications use on a daily basis will be reviewed on a case-by-case basis. Patients may be excluded if medical therapies could interfere with the study endpoints.
8. Patients will be excluded if they have an uncontrolled seizure disorder.
9. Patients on miglustat at the start of the study will be excluded if the dose of miglustat cannot be held constant for the duration of the study. The miglustat dose must have been constant for two months prior to the baseline NIH evaluation. Patients will be withdrawn if they initiate miglustat use after entering the study.
10. Patient who are at risk for gastric hemorrhage (preexisting esophageal varices or peptic ulcer disease).
11. Patients on a sodium restricted diet for medical reasons.
12. The following laboratory test abnormalities will exclude patients from the study:

    * a. AST or ALT elevated greater than 4-fold upper limit of normal. Note: NPC patients frequently have transaminase levels 2-3 fold above normal.
    * b. Anemia defined as two standard deviations below normal for age and gender.
    * c. Platelet count less than 75,000.
    * d. Elevated serum creatine level
    * e. Hematuria or proteinuria

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Vanier MT, Millat G. Niemann-Pick disease type C. Clin Genet. 2003 Oct;64(4):269-81. doi: 10.1034/j.1399-0004.2003.00147.x. PMID 12974729
- [Background] Carstea ED, Morris JA, Coleman KG, Loftus SK, Zhang D, Cummings C, Gu J, Rosenfeld MA, Pavan WJ, Krizman DB, Nagle J, Polymeropoulos MH, Sturley SL, Ioannou YA, Higgins ME, Comly M, Cooney A, Brown A, Kaneski CR, Blanchette-Mackie EJ, Dwyer NK, Neufeld EB, Chang TY, Liscum L, Strauss JF 3rd, Ohno K, Zeigler M, Carmi R, Sokol J, Markie D, O'Neill RR, van Diggelen OP, Elleder M, Patterson MC, Brady RO, Vanier MT, Pentchev PG, Tagle DA. Niemann-Pick C1 disease gene: homology to mediators of cholesterol homeostasis. Science. 1997 Jul 11;277(5323):228-31. doi: 10.1126/science.277.5323.228. PMID 9211849
- [Background] Naureckiene S, Sleat DE, Lackland H, Fensom A, Vanier MT, Wattiaux R, Jadot M, Lobel P. Identification of HE1 as the second gene of Niemann-Pick C disease. Science. 2000 Dec 22;290(5500):2298-301. doi: 10.1126/science.290.5500.2298. PMID 11125141
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-CH-0185.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Phase A/NAC Phase B: These patients were randomized to receive the placebo in Phase A and study drug (NAC) in Phase B of the trial
- NAC Phase A/Placebo Phase B: These patients were randomized to receive study drug (NAC) in Phase A and placebo in Phase B
Period: Overall Study
Arm/Group | Placebo Phase A/NAC Phase B | NAC Phase A/Placebo Phase B
Started | 17 | 18
Completed | 15 | 15
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Phase A/NAC Phase B | NAC Phase A/Placebo Phase B | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 13 | 25
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34
  Costa Rica | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Oxysterol Levels
Time Frame: Six months
Population: Every patient in the trial received the study drug as well as the placebo.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | NAC Phase | Placebo Phase
Number analyzed (Participants) | 30 | 30
ng/mL | 28.09 (2.152) | 27.64 (2.045)

ADVERSE EVENTS:
Arm/Group | Placebo Phase A/NAC Phase B | NAC Phase A/Placebo Phase B
Serious Adverse Events (participants affected / at risk) | 3/17 | 5/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Phase A/NAC Phase B (N=17) | NAC Phase A/Placebo Phase B (N=18)
Elevated Liver Enzymes (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hospitalization for seizure (Nervous system disorders) | 1 (1) | 2 (2) — Unanticipated hospitalization
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decreased blood counts (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes